CLINICAL TRIAL: NCT00257868
Title: Rivastigmine for the Prevention of Postoperative Delirium After Cardiac Surgery
Brief Title: Rivastigmine for the Prevention of Postoperative Delirium in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EKBB 204/05; CENA713CCH01
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-07

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

INTERVENTIONS:
Drug: Rivastigmine prevention of delirium

SUMMARY:
The purpose of this study is to determine whether Rivastigmine is effective for the prevention of postoperative delirium in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Postoperative delirium is a frequent complication after cardiac surgery. In the literature an incidence ranging from 0 - 72 % is reported. The aetiology of this complication is multifactorial. A decline in cerebral cholinergic transmission as well as perioperative cerebral hypoperfusion or a systemic inflammatory response triggered by the extracorporeal circulation have been suspected. Advanced age is the most important patient-related risk factor. A perioperative delirium is an extremely unpleasant experience for the affected patients. Equally important is the fact that a delirium is associated with a prolonged length of stay on the intensive care unit and in hospital. Furthermore, patients who develop delirium have an increased six-month mortality. Recently successful treatment and prevention of the delirium with cholinesterase inhibitors such as rivastigmine have been reported.

The proposed study will test the hypothesis that prophylactically administered rivastigmine is able to prevent or at least reduce the symptoms of the postoperative delirium in elderly patients undergoing elective cardiac surgery with extracorporeal circulation.

This study is designed as a double blind randomised placebo controlled trial. Half the patients will receive placebo. The other half will receive rivastigmine 1.5m-1.5mg-1.5mg (oral solution), starting on the evening preceding the operation and for the first seven days postoperatively. Patients in both groups who develop delirium will be treated with a rescue medication consisting of lorazepam and haloperidol.

Measurements will include the incidence of delirium assessed using the Confusion Assessment Method (CAM). The severity of symptoms will by characterised by the Mini Mental Score and clock drawing. Further measurements will include the prescribed doses of rescue medication, the length of stay on intensive care and in hospital, the time of extracorporeal circulation, and laboratory parameters such as CRP, albumin, lymphocyte count, vitamin B12 and folic acid levels. Side effects of rivastigmine will be quantified.

The primary endpoint of this study is the incidence of delirium. Secondary endpoints will be the severity of delirium, the used doses of rescue medication, and length of stay (intensive care and hospital).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery with use of extracorporeal circulation
* Aged 65 or more

Exclusion Criteria:

* "redo" procedures
* anticipated use of succinylcholine during operation
* contraindications to rivastigmine
* preoperative mini mental score < 15

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-01; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Development of postoperative delirium within 7 days after cardiac surgery

SECONDARY OUTCOMES:
Severity of delirium occurring within 7 days after cardiac surgery
Length of stay (intensive care and hospital)
Amount of drugs used for rescue therapy of delirium

CONTACTS AND LOCATIONS:
Overall Officials: Luzius A Steiner, MD PhD, Principal Investigator — Department of Anaesthesia, University Hospital Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland